CLINICAL TRIAL: NCT05658991
Title: Retinal Functional Changes With Different Dietary Habits.
Brief Title: Electrophysiological Changes With Diet.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Assistant professor of Ophthalmology, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC-12.2022
Record Dates: First submitted 2022-12-11; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Fasting, Intermittent; Fasting Hypoglycemia; Fasting; Obesity; Diabetes
Keywords: Fasting; Ramadan; Diet; Retina; Electroretinogram
MeSH Terms: conditions — Intermittent Fasting; Hypoglycemia; Fasting; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent fasting healthy group (Active Comparator): Healthy participants with intermittent fasting dietary habit.
  Interventions: Diagnostic Test: Retinal electrophysiology
- Obesity group (Active Comparator): Subjects with body mass index more than 30.
  Interventions: Diagnostic Test: Retinal electrophysiology

INTERVENTIONS:
Diagnostic Test: Retinal electrophysiology — Retinal electrophysiology to assess retinal function before and with fasting during ramadan in both groups.

SUMMARY:
Dietary habits may affect our body by certain mechanisms, visual sense is one of the most vital human senses that needs special attention in our daily habits.

DETAILED DESCRIPTION:
Retinal function directly related to our quality of vision, different drugs can affect our vision in certain ways, however, out unhealthy dietary habits can indirectly affect our quality of life and vision.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects with intermittent fasting.
* obese subjects with body mass index more than 30.

Exclusion Criteria:

* patients with any retinal diseases that may ter retinal functional test.
* patients on systemic drugs that may alter retinal function.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-11 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Retinal function amplitude | Baseline and one month after fasting in both groups.
  Changes in amplitude of retinal electrophysiology in both groups measured in nano volt/degree.

SECONDARY OUTCOMES:
Retinal function latency. | Baseline and one month after fasting in both groups.
  Changes in latency of retinal electrophysiology in both groups measured in milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Tabl, MD, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy Tabl, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: No